CLINICAL TRIAL: NCT06836791
Title: Topical 15% Trichloroacetic Acid Versus Silver Nitrate Cauterization in the Management of Idiopathic Childhood Epistaxis: A Prospective Double-Blinded, Randomized Clinical Trial
Acronym: Epistaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youssef Zaki (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Sponsor-Investigator, Youssef Zaki, principal investigator, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200
Record Dates: First submitted 2025-01-29; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Anterior Epistaxis
MeSH Terms: interventions — Silver Nitrate; Trichloroacetic Acid

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, double-blinded study that was held at our tertiary referral center, Otorhinolaryngology Department, Kafrelsheikh University, Egypt.
  All patients' parents or assigned caregivers signed written informed consent for participation in this trial. Patients who sought help complaining of recurrent epistaxis episodes either with or without active bleeding at the time of presentation were invited to participate in the study. All patients aged between 4 and 16 years with at least once weekly in the last 4 weeks with visible anterior bleeding sources either unilateral or bilateral from Little's area were included in the study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver nitrate group (Experimental): All procedures were performed as office-based procedures under the influence of local anesthesia.
  Group (A) Silver nitrate group: Patients were treated with silver nitrate chemical cauterization. Prior to cauterization, 2 cotton packs soaked in 10% lignocaine spray were introduced into each nostril for 5-10 minutes. Then, a cotton-tipped applicator dipped in 25% silver nitrate solution was applied to the bleeding point, and the sample was firmly pressed for 1 minute. In the case of bleeding, a second application of silver nitrate solution was applied to the area, after which a cotton tip applicator was applied to the area for 30 s with cauterization of all the feeding blood vessels around the bleeding point. This was followed by the prescription of an antiseptic soothing cream topically twice daily for 2 weeks.
  Interventions: Procedure: chemical cautrizating agents to stop epistaxis; Drug: Silver Nitrate
- Trichloroacetic acid group (Experimental): Group (B) The TCA group: Patients underwent chemical cauterization with 15% TCA solution via the same technique. If there was active nasal bleeding, prior to cauterization, a cotton pack soaked in a nasal decongestant such as oxymetazoline or a 10% lignocaine spray was introduced into the nostril for 5-10 minutes. Patients were offered topical antiseptics for two weeks. Both groups were offered analgesics according to their condition.
  Interventions: Procedure: chemical cautrizating agents to stop epistaxis; Drug: Trichloroacetic Acid Topical

INTERVENTIONS:
Procedure: chemical cautrizating agents to stop epistaxis — All procedures were performed as office-based procedures under the influence of local anesthesia.Patients were treated with chemical cauterization. Prior to cauterization, 2 cotton packs soaked in 10% lignocaine spray were introduced into each nostril for 5-10 minutes. Then, a cotton-tipped applicator dipped in chemical cautrizating agents solution was applied to the bleeding point, and the sample was firmly pressed for 1 minute. In the case of bleeding, a second application of chemical cautrizating agents solution was applied to the area, after which a cotton tip applicator was applied to the area for 30 s with cauterization of all the feeding blood vessels around the bleeding point. This was followed by the prescription of an antiseptic soothing cream topically twice daily for 2 weeks.
Drug: Silver Nitrate — silver nitrate is chemical cautrizing agent ,in the study ,the investigators use it in treatment of anterior epistaxis in children by dissolving silver nitrate crystals in normal saline solution before using.
  Arms: Silver nitrate group
Drug: Trichloroacetic Acid Topical — trichloroacetic acid is well known peeling agent ,in the study the investigators use it as chemical cautrizing agent to treat anterior epistaxis in children .
  Other Names: TCA
  Arms: Trichloroacetic acid group

SUMMARY:
the invistigators aim to explore the efficacy of trichloroacetic acid as a chemical cauterization agent and compare it with that of silver nitrate in the treatment of idiopathic epistaxis in children.

DETAILED DESCRIPTION:
Epistaxis is a very distressing complaint in otorhinolaryngology that affects nearly 10-12% of the population worldwide . Epistaxis in children is even more common. Approximately half of the children had one or more episodes of epistaxis by the age of 10 .

The source of epistaxis may be anterior or posterior; in children, epistaxis is commonly anterior, originating mainly from the anterior part of the nasal septum called Little's area, in which a confluence of veins named Kiesselbach's plexus is the main area to blame . Anterior epistaxis is commonly related to local trauma, such as nose picking or crust formation, or local inflammation, such as upper airway infection and vestibulitis, due to bacterial inhabitants that lead to crusting and precipitation of epistaxis episodes.

In the literature, there are various modalities for the treatment of anterior epistaxis, such as nose pinching and anterior nasal packing in emergent cases and medical treatment in between attacks, which are considered first aid, and whenever they fail, we shift to alternative methods that are considered invasive but more effective .

One of the currently utilized modalities that has been shown to be effective in the management of epistaxis is chemical cauterization of the prominent vessels in Little's area . In 1932, Little was the first to introduce the idea of using silver nitrate as a chemical cautery agent in the treatment of anterior epistaxis, which results in coagulation of bleeding vessels and tissue destruction .

Another option for chemical cauterization is trichloroacetic acid (TCA), which causes protein denaturation . Trichloroacetic acid is available, inexpensive, and easy to use as a chemical cautery solution. However, there is not yet adequate evidence in the literature for the use of TCA in the treatment of epistaxis.

Therefore, the invistigators aimed to explore the efficacy of trichloroacetic acid as a chemical cauterization agent and compare it with that of silver nitrate in the treatment of idiopathic epistaxis in children.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged between 4 and 16 years at least once weekly in the last 4 weeks with visible anterior bleeding sources either unilateral or bilateral from Little's area were included in the study.

Exclusion Criteria:

* All patients with documented coagulopathy, those with sinonasal or nasopharyngeal masses, those with active rhinosinusitis or severe allergic rhinitis or severe septal deviation

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
rebleeding from the nose | 12 weeks
  Patients were followed at regular visits at the 1st, 2nd, 4th, and 12th week intervals.
  The main outcomes after chemical cauterization were rebleeding from the nose if present during or after the procedure. The success of post chemical cauterization was assessed through the complete cessation of epistaxis. Patients with reported recurrence of bleeding from the nose within 12 weeks of intervention were considered to have failed. rebleeding assessed according to number of bleeds and severity of the attacks.

SECONDARY OUTCOMES:
pain after procedure | 7 days after caurication
  Pain was assessed via the Wong-Baker FACES® Pain Rating Scale [9], which is represented by a series of faces ranging from 0 (smiling face) to 10 (crying face), with 10 referring to the most intense pain. Following a brief explanation, the child can select the face that best represents. We asked the parents to fill out the questionnaire by asking their children to point out the suitable face by the third day postintervention and then reporting it at their 1st-week visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafrelsheikh, Kafrelsheikh, Egypt